CLINICAL TRIAL: NCT05162261
Title: A Randomized, Masked (Evaluator), Controlled, Prospective Study Evaluating the Effectiveness and Safety of the Tixel® Medical Device, Versus LipiFlow® in the Treatment of Meibomian Gland Dysfunction
Brief Title: to Evaluate the Effectiveness and Safety of the Tixel® , VS LipiFlow® in the Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN 0858
Record Dates: First submitted 2021-11-21; First posted 2021-12-17 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Syndromes; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A Randomized, Masked (Evaluator), Controlled, Prospective, open label study.
Who Masked: Outcomes Assessor
Masking Description: Blinded Evaluator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tixel Group (Experimental): Screening and baseline visits, Treatment- 3 treatment sessions, followed by 2 Follow up sessions, 1and 3 months after the last treatment visit. Subject will be questioned about Discomfort and Pain Questionnaires (self-assessed) and OSDI questionnaire.
  Interventions: Device: Tixel C
- LipiFlow (Active Comparator): LipiFlow: Screening and baseline visits,Treatment session, followed by 2 Follow up sessions, 1and 3 months after the last treatment visit. Subject will be questioned about Discomfort and Pain Questionnaires (self-assessed) and OSDI questionnaire.
  Interventions: Device: LipiFlow

INTERVENTIONS:
Device: Tixel C — Tixel C by Novoxel®, Israel is a thermomechanical system developed for fractional treatment. The system is designed for the treatment of soft tissue by direct conduction of heat, enabling tissue coagulation combined with micro ablation with low thermal damage to the surrounding tissue.
  Arms: Tixel Group
Device: LipiFlow — Thermal pulsation (LipiFlow) consists of the localized application of heat and therapeutic pressure on the four eyelids (upper and lower) with the aim of improving drainage of the Meibomian glands.
  Arms: LipiFlow

SUMMARY:
A Randomized, Masked (Evaluator), Controlled, Prospective Study Evaluating the Effectiveness and Safety of the Tixel® Medical Device, Versus LipiFlow® in the Treatment of Meibomian Gland Dysfunction

DETAILED DESCRIPTION:
Randomized, open-label study comparing the Tixel device to LipiFlow System. Up to 110 patients (220 eyes) to be randomized in up to 5 clinical sites in the United States.

Evaluators will be masked as to the randomization assignments. Both eyes will receive the same randomized assignment and both eyes of each patient will be evaluated at all time points.

Data from both eyes will be using in the statistical analysis. The random-effects model adjusts the standard error (SE) and the confidence interval (CI) for within-person correlation between eyes.

Protocol Rev. 7.0 update: Addition of protocol extension to the current protocol: stage 1- main protocol for all patients and stage 2- extension protocol to a sub-group of patients only in the Tixel arm for additional follow-up visit 6 months post last treatment.

ELIGIBILITY:
Main Study (Stage1) Inclusion Criteria:

1. Age 22 years and older of any gender or race.
2. Provision of written informed consent prior to study participation.
3. Willingness and ability to return for all study visits.
4. Reports dry eye symptoms for three months prior to the study.
5. Ocular Surface Disease Index (OSDI) score between 23-79.
6. Tear break-up time (TBUT) <10 seconds in both eyes.
7. Agreement/ability to abstain from dry eye/MGD medications for the time between the treatment visit/s and the final study visit. Ocular lubricants are allowed if no changes are made during the study.
8. Reports having to use artificial tears or lubricants regulatory over the past month to relieve dry eye symptoms.
9. Meibomian gland obstruction in both eyes based on a total Meibomian Gland Secretion Score ≤12 in each eye.
10. At least 15 glands in each lower eyelid should be expressible, with a sterile cotton swab, at the slit lamp.

Main Study (Stage1) Exclusion Criteria:

1. History of ocular surgery including intraocular, oculo-plastic, corneal or refractive surgery within 6 months.
2. Patient with giant papillary conjunctivitis.
3. Patient with punctal plugs or who have had punctal cautery.
4. Ocular injury or trauma, chemical burns, or limbal stem cell deficiency within 3 months of the baseline examination.
5. Active ocular herpes zoster or simplex of eye or eyelid or a history of these any time.
6. Patient who are aphakic.
7. Cicatricial lid margin disease identified via slit lamp examination, including pemphigoid, symblepharon, etc.
8. Active ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac, or eyelids including a hordeolum or stye).
9. Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months (e.g., retinitis, macular inflammation, choroiditis, uveitis, iritis, scleritis, episcleritis, keratitis).
10. Ocular surface abnormality that may compromise corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy).
11. Lid surface abnormalities (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis) that affect lid function in either eye.
12. Anterior blepharitis (staphylococcal, demodex or seborrheic grade 3 or 4).
13. Systemic disease conditions that cause dry eye (e.g., Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, Sjogren's syndrome).
14. Use of any of the following medications:

    1. Systemic medication(s) that is known to cause ocular dryness (e.g. antihistamine, diuretics, anti-hypertensives, anti-depressants, hormone therapy) whose dose of this medication(s) has not been stable within 30 days prior to enrolment. There must be no anticipated adjustments to the dose of these medications for the duration of the trial;
    2. Oral tetracyclines or azithromycin within 30 days prior to enrolment; or
    3. Topical anti-glaucoma medications within 30 days prior to enrolment.
    4. Any other systemic medication as per to the Investigator's discretion.
15. Women in childbearing age who are pregnant, nursing, or not utilizing adequate birth control measures.
16. Individuals using isotretinoin (Accutane) within 1 year, cyclosporine-A (Restasis) or lifitegrast ophthalmic solution (Xiidra) within 45 days prior to study treatment (day 0), or any other dry eye or MGD medications (antibiotics, non-steroidal anti-inflammatory drugs, corticosteroids) for at least 2 weeks and to maintain abstinence throughout the duration of the study (ocular lubricants are allowed if no changes are made during the study).
17. Individuals wearing contact lenses 1 month prior study treatment (day 0), and at any point during the study.
18. Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
19. An impaired immune system condition or use of immunosuppressive medication.
20. Collagen disorders, keloid formation and/or abnormal wound healing.
21. Previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans for such treatment during the course treatment, or before complete healing of such treatments has occurred.
22. Any patient who takes or has taken any oral or topical medications, such as but not limited to topical retinoid (e.g., Retin-A), chemical peels, Latisse, Lash Boost which may cause fragile skin or impaired skin healing in the treatment area during the last 3 months and in the entire study period.
23. Any patient who has a history of bleeding coagulopathies.
24. Any patient who has tattoos or permanent makeup in the treated area.
25. Any patient who has burned, blistered, irritated, or sensitive skin in any of the areas to be treated.
26. Individuals using another ophthalmic investigational device or agent within 30 days of study participation.
27. Any of the following dry eye treatments:

    1. Office-based dry eye treatment (e.g. IPL, LipiFlow, iLux, TearCare, Tixel, etc.) within 12 months prior to enrolment;
    2. Meibomian gland expression within 6 months prior to enrolment;
    3. Blephex or debridement within 3 months prior to enrollment is an exclusion;
    4. Punctal occlusion or punctal plug placement within 30 days prior to enrolment;
    5. Use of iTear or TrueTear device within the past 2 weeks. (Subjects must refrain from using these devices for the duration of the study.); or
    6. Any history of meibomian gland probing
28. Use of at-home warm compresses or lid hygiene products while participating in study.
29. IOP higher than 19 mmHg.
30. Use of Botulinum-Toxin in the last 6 months prior to the treatment in the treatment area.
31. Any co-existing condition, either ocular or non-ocular that, in the judgement of the investigator, could affect the safety or effectiveness of treatment or the compliance of the subject to the protocol.

Study Extension (Stage 2)- Inclusion Criteria

* Subjects who have completed the main study CLN 0858 (stage 1) in the Tixel arm.
* TBUT -change from baseline in 1-month FU or 3-months FU was 2.5 seconds or above at least in one eye in the main study.
* Provision of written informed consent for stage 2.
* Agreement/ability to abstain from dry eye/MGD medications for the time in the extension study. Ocular lubricants are allowed if no changes are made during the study.

Study Extension (Stage 2)-Exclusion Criteria

* Same as in the main study (stage 1).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Berdy, MD, Principal Investigator — Ophthalmology Associates 12990 Manchester Rd., Ste. 200 St. Louis, MO 63131 314-966-3377
Locations (5):
- United States (5):
  - Gordon Schanzlin New Vision Institute, La Jolla, California
  - Visionary Research Institute, Newport Beach, California
  - Moyes Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - PNV Clinical Research, LLC, Texas City, Texas

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Tixel Group | LipiFlow
Started | 54; 108 Eyes | 55; 110 Eyes
Completed | 45; 90 Eyes | 53; 106 Eyes
Not Completed | 9; 18 Eyes | 2; 4 Eyes

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized subjects. Subjects were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tixel Group | LipiFlow | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.4) | 61.7 (12.8) | 61.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 49 | 50 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 50 | 51 | 101
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 55 | 109
Ftzpatrick skin type [Count of Participants; unit: Participants] — Assessment of subject's skin color was determined prior to study procedure by the Investigator using the FSS. The scale delineates skin color into the categories as shown below :
  Skin Type Description Type I White skin that never tans and always burns easily Type II White skin that tans slightly and always burns easily Type III Light brown skin that tans gradually and can burn moderately Type IV Moderately brown skin that tans well and burns slightly Type V Dark brown skin that tans profusely and burns rarely Type VI Black skin with deep pigmentation that never burns
  Participants
    Type 1 | 1 | 1 | 2
    Type 2 | 18 | 17 | 35
    Type 3 | 15 | 21 | 36
    Type 4 | 16 | 13 | 29
    Type 5 | 3 | 2 | 5
    Type 6 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Changes in Tear Break Up Times (TBUT) to the 4-weeks Follow-up Exam
Description: Change from baseline to the 4-weeks follow-up exam in Tear Break Up Times (TBUT), as assessed by a masked rater.
  TBUT - Tear Break-Up Time, is a clinical test used to evaluate the stability of the tear film on the surface of the eye. It measures the time it takes for dry spots to appear on the cornea after a blink. A shorter TBUT indicates a more unstable tear film, which can be a sign of dry eye disease or other ocular surface disorders.
  Tear Break-Up Time (TBUT) is typically scored by the time (in seconds). The general interpretation of TBUT scores is as follows:
  Normal TBUT: More than 10 seconds Borderline TBUT: 5 to 10 seconds Abnormal/Low TBUT: Less than 5 seconds
Time Frame: Tixel arm: Baseline and 4 weeks after last treatment (8 weeks post baseline). LipiFlow arm: Baseline and 4 weeks after treatment (4 weeks post baseline).
Population: 48 Tixel subjects and 52 LipiFlow subjects completed the Baseline and 4-week FU TBUT examination.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 48 | 52
Number analyzed (Eyes) | 96 | 104
seconds
  Baseline | 4.3 (1.5) | 4.6 (1.8)
  change from baseline - 4 weeks FU | 3.0 (3.2) | 2.7 (2.7)

2. Primary Outcome: Comparison of the Incidence of Device-related Ocular Adverse Events
Description: Comparison of the incidence of device-related Ocular adverse events for the two treatment arms
Time Frame: Tixel arm: Baseline to 12 weeks after last treatment (16 weeks post baseline). LipiFlow arm: Baseline to 12 weeks after treatment (12 weeks post baseline).
Population: Safety Population: Included all subjects who were treated. All safety analyses were performed using the Safety population
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 53 | 53
Number analyzed (Eyes) | 106 | 106
participants | 0 | 0

3. Secondary Outcome: Changes in Patient OSDI
Description: Change from baseline in patient symptoms using Ocular Surface Disease Index (OSDI) at 4-weeks and 12-weeks follow-up exam.
  The Ocular Surface Disease Index (OSDI) is a questionnaire designed to assess the severity of dry eye disease.
  OSDI Questionnaire
  The questionnaire consists of 12 questions divided into three subscales:
  Ocular Symptoms Visual Functioning Environmental Triggers
  Scoring System
  The scoring for the OSDI is based on a scale from 0 to 100, where higher scores indicate more severe symptoms. Each question is scored as follows:
  0: None of the time
  1. Some of the time
  2. Half of the time
  3. Most of the time
  4. All of the time
  Interpretation of OSDI Scores
  The OSDI scores are generally interpreted as follows:
  0-12: Normal or no dry eye 13-22: Mild dry eye 23-32: Moderate dry eye 33-100: Severe dry eye
Time Frame: as for outcome 2
Population: Per Protocol (PP) Population: Included all subjects who completed all study treatments as randomized, completed the 4-week follow-up visit, and who had no major protocol deviations. The PP population was used for the effectiveness endpoint analyses.Tixel subects and lipiflow subjects completed baseline, 4 weeks OSDI and 12 weeks OSDI.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 48 | 52
Number analyzed (Eyes) | 96 | 104
score on a scale
  Baseline | 50.2 (18.3) | 49.4 (15.5)
  Change 1 month - Baseline | -26.4 (21.1) | -18.8 (21.0)
  Change 3 months - Baseline: number analyzed (Participants) | 45 | 52
  Change 3 months - Baseline: number analyzed (Eyes) | 90 | 104
  Change 3 months - Baseline | -28.6 (22.4) | -21.9 (18.5)

4. Secondary Outcome: Changes in Tear Break Up Times (TBUT) to the 12-weeks Follow-up Exam
Description: Changes from baseline to the 12-weeks follow-up exam in Tear Break Up Times (TBUT), as assessed by a masked rater.
  BUT - Tear Break-Up Time, is a clinical test used to evaluate the stability of the tear film on the surface of the eye. It measures the time it takes for dry spots to appear on the cornea after a blink. A shorter TBUT indicates a more unstable tear film, which can be a sign of dry eye disease or other ocular surface disorders.
  Tear Break-Up Time (TBUT) is typically scored by the time (in seconds). The general interpretation of TBUT scores is as follows:
  Normal TBUT: More than 10 seconds Borderline TBUT: 5 to 10 seconds Abnormal/Low TBUT: Less than 5 seconds
Time Frame: Tixel arm: Baseline and 12 weeks after last treatment (16 weeks post baseline). LipiFlow arm: Baseline and 12 weeks after treatment (12 weeks post baseline).
Population: Per Protocol (PP) Population: Included all subjects who completed all study treatments as randomized, completed the 4-week follow-up visit, and who had no major protocol deviations. The PP population was used for the effectiveness endpoint analyses.
Measure: Median (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 45 | 52
Number analyzed (Eyes) | 90 | 104
seconds
  Baseline | 4.3 (1.5) | 4.6 (1.8)
  TBUT change from baseline to 12 weeks FU | 3.1 (4.3) | 3.3 (3.6)

5. Secondary Outcome: Changes in MGS to 4-weeks and 12-weeks Follow-up Exam
Description: score on a scale at baseline, 4-weeks and 12-weeks follow-up exam in Meibomian Gland (MGS), as assessed by a masked rater.
  The Meibomian Gland Score (MGS) is a clinical tool used to evaluate the function of the meibomian glands.
  Scoring Criteria
  Each gland is assessed and scored based on the quality of the expressed secretion:
  0: No secretion
  1. Inspissated
  2. Cloudy
  3. Clear liquid
  Interpretation of MGS Minimal MGS score = 0 in each eye (15 glands evaluated in each eye) Maximal MGS score = 45 in each eye (15 glands evaluated in each eye) Low MGS: (below 12) Indicates poor function or obstruction of the meibomian glands, suggesting MGD.
Time Frame: as for outcome 2
Population: Per Protocol (PP) Population: Included all subjects who completed all study treatments as randomized, completed the 4-week follow-up visit, and who had no major protocol deviations. The PP population was used for the effectiveness endpoint analyses. subject in the tixel group and subject in the lipiflow group comparisoon at baseline, 4 weeks and 12 weeks visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 48 | 52
Number analyzed (Eyes) | 96 | 104
score on a scale
  Baeline | 7.2 (2.5) | 7.4 (2.6)
  Change 1 Month- Baseline | 9.0 (10.4) | 7.3 (8.8)
  Change 3 Months - Baseline: number analyzed (Participants) | 45 | 52
  Change 3 Months - Baseline: number analyzed (Eyes) | 90 | 104
  Change 3 Months - Baseline | 11.3 (11.4) | 10.5 (12.2)

6. Secondary Outcome: Score on a Scale During Treatment Discomfort and Pain Questionnaires (Each Self-assessed by VAS)
Description: Discomfort and Pain from the treatment (Tixel or LipiFlow) using the questionnaires assessed by the subject. These are visual analogue scale (VAS) questionnaires using a scale from 0-10 to assess eye discomfort and pain. Both questionnaires are to be self-assessed by the patient immediately following treatment.
  Interpetation for the assessment:
  score 0- no discomfort / pain score 5 - moderate discomfort / pain score 10 - worst possible discomfort / pain
Time Frame: Tixel arm: 4 weeks (treatment 1- day 0, treatment 2- 2 weeks, treatment 3- 4 weeks). LipiFlow arm: On treatment day - day 0 (only one treatment for this arm)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 53 | 53
Number analyzed (Eyes) | 106 | 106
score on a scale
  Discomfort Treatment 1 -OD: number analyzed (Eyes) | 53 | 53
  Discomfort Treatment 1 -OD | 2.8 (1.9) | 1.5 (1.6)
  Discomfort Treatment 1 -OS: number analyzed (Eyes) | 53 | 53
  Discomfort Treatment 1 -OS | 2.6 (1.8) | 1.7 (2.1)
  Discomfort Treatment 2 - OD: number analyzed (Participants) | 50 | 0
  Discomfort Treatment 2 - OD: number analyzed (Eyes) | 50 | 0
  Discomfort Treatment 2 - OD | 2.7 (1.8) |
  Discomfort Treatment 2 - OS: number analyzed (Participants) | 50 | 0
  Discomfort Treatment 2 - OS: number analyzed (Eyes) | 50 | 0
  Discomfort Treatment 2 - OS | 2.6 (1.7) |
  Discomfort treatment 3 -OD: number analyzed (Participants) | 50 | 0
  Discomfort treatment 3 -OD: number analyzed (Eyes) | 50 | 0
  Discomfort treatment 3 -OD | 2.5 (2.0) |
  Discomfort treatment 3 -OS: number analyzed (Participants) | 50 | 0
  Discomfort treatment 3 -OS: number analyzed (Eyes) | 50 | 0
  Discomfort treatment 3 -OS | 2.5 (2.0) |
  Pain- Treatment 1 -OD: number analyzed (Eyes) | 53 | 53
  Pain- Treatment 1 -OD | 2.5 (1.9) | 0.8 (1.2)
  Pain- Treatment 1-OS: number analyzed (Eyes) | 53 | 53
  Pain- Treatment 1-OS | 2.5 (1.9) | 0.9 (1.5)
  Pain - Treatment 2 -OD: number analyzed (Participants) | 50 | 0
  Pain - Treatment 2 -OD: number analyzed (Eyes) | 50 | 0
  Pain - Treatment 2 -OD | 2.5 (1.9) |
  Pain - Treatment 2- OS: number analyzed (Participants) | 50 | 0
  Pain - Treatment 2- OS: number analyzed (Eyes) | 50 | 0
  Pain - Treatment 2- OS | 2.3 (1.8) |
  Pain - Treatment 3 -OD: number analyzed (Participants) | 50 | 0
  Pain - Treatment 3 -OD: number analyzed (Eyes) | 50 | 0
  Pain - Treatment 3 -OD | 2.2 (2.0) |
  Pain - Treatment 3 -OS: number analyzed (Participants) | 50 | 0
  Pain - Treatment 3 -OS: number analyzed (Eyes) | 50 | 0
  Pain - Treatment 3 -OS | 2.2 (1.9) |

7. Secondary Outcome: Corneal Fluorescein Staining Slit Lamp Evaluation Scores and Change From Baseline
Description: Changes from baseline following treatment for the test and control devices for the following assessments:
  Ocular Surface Staining (to evaluate the integrity of the corneal epithelium by identifying areas of damage or staining)
  Grading scale:
  0 = Normal - No staining
  1. = Mild - Superficial stippling micropunctate staining
  2. = Moderate - Macropunctate staining with some coalescent areas
  3. = Severe - Numerous coalescent macropunctate areas and/or patches
  5 regions (superior, temporal, central, nasal, and inferior) are graded for each eye. total score range from 0 -15.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 53 | 53
Number analyzed (Eyes) | 106 | 106
score on a scale
  Baseline | 3.1 (2.4) | 2.9 (2.2)
  Post Treatment 1 | 2.1 (2.1) | 2.0 (1.9)
  Post Treatment 2: number analyzed (Participants) | 50 | 0
  Post Treatment 2: number analyzed (Eyes) | 100 | 0
  Post Treatment 2 | 1.4 (1.6) |
  Post Treatment 3: number analyzed (Participants) | 50 | 0
  Post Treatment 3: number analyzed (Eyes) | 100 | 0
  Post Treatment 3 | 0.9 (1.3) |
  1 Month Follow-up: number analyzed (Participants) | 48 | 52
  1 Month Follow-up: number analyzed (Eyes) | 96 | 104
  1 Month Follow-up | 1.2 (1.9) | 1.5 (1.6)
  3 Months Follow up: number analyzed (Participants) | 45 | 53
  3 Months Follow up: number analyzed (Eyes) | 90 | 106
  3 Months Follow up | 1.3 (2.2) | 1.3 (1.8)
  Change 1 Month - Baseline: number analyzed (Participants) | 48 | 52
  Change 1 Month - Baseline: number analyzed (Eyes) | 96 | 104
  Change 1 Month - Baseline | -1.9 (2.3) | -1.4 (2.2)
  Change 3 Months - Baseline: number analyzed (Participants) | 45 | 53
  Change 3 Months - Baseline: number analyzed (Eyes) | 90 | 106
  Change 3 Months - Baseline | -1.7 (2.3) | -1.6 (2.1)

8. Secondary Outcome: The Mean Changes From Baseline in IOP for All Eyes on the Tixel and Lipiflow Arms
Description: Changes from baseline following treatment for the test and control devices for:
  Intraocular Pressure
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 53 | 53
Number analyzed (Eyes) | 106 | 106
score on a scale
  Baseline | 13.3 (2.4) | 13.5 (2.8)
  Change in IOP (mmHG) from Baseline to 1 month follow up: number analyzed (Participants) | 48 | 52
  Change in IOP (mmHG) from Baseline to 1 month follow up: number analyzed (Eyes) | 96 | 104
  Change in IOP (mmHG) from Baseline to 1 month follow up | 0.4 (2.5) | 0.2 (2.5)
  change in IOP (mmHG) from Baseline to 3 months follow up: number analyzed (Participants) | 45 | 53
  change in IOP (mmHG) from Baseline to 3 months follow up: number analyzed (Eyes) | 90 | 106
  change in IOP (mmHG) from Baseline to 3 months follow up | 0.1 (2.7) | 0.3 (2.4)

9. Secondary Outcome: Ocular Surface Conjunctival Lissamine Green Staining Changes From Baseline
Description: Changes from baseline following treatment for the test and control devices for the following assessments:
  Lissamine staining scores (to assess the health of the conjunctival and corneal epithelium, particularly in dry eye disease, by identifying areas of damaged or dead cells).
  Grading scale:
  0 = Normal - No staining
  1. = Mild - Superficial stippling micropunctate staining
  2. = Moderate - Macropunctate staining with some coalescent areas
  3. = Severe - Numerous coalescent macropunctate areas and/or patches
  6 regions (nasal, superior nasal, inferior nasal, temporal, superior temporal, inferior temporal) are graded for each eye. The total score range for each eye is 0-18.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 53 | 53
Number analyzed (Eyes) | 106 | 106
score on a scale
  Basline | 2.4 (2.8) | 2.4 (2.5)
  Change from baseline to 1 month FU: number analyzed (Participants) | 48 | 52
  Change from baseline to 1 month FU: number analyzed (Eyes) | 96 | 104
  Change from baseline to 1 month FU | -0.9 (2.3) | -1.2 (2.7)
  Change from baseline to 3 months FU: number analyzed (Participants) | 45 | 53
  Change from baseline to 3 months FU: number analyzed (Eyes) | 90 | 106
  Change from baseline to 3 months FU | -1.3 (2.7) | -1.2 (3.0)

10. Other Pre Specified Outcome: Extension Study Endpoint 1
Description: Durability of the clinical benefit effect at 6-months FU visit assessed by OSDI parameter for a Tixel sub-group population only.
Time Frame: Baseline and 6 months post-last treatment (7 months post-baseline)
Population: Tixel sub-group population
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
score on a scale
  Baseline | 46.2 (19.7)
  6 months FU visit | 21.9 (19.4)
  6 months FU score change from baseline | -24.3 (26.5)

11. Other Pre Specified Outcome: Extension Study Endpoint 2
Description: Durability of the clinical benefit effect at 6-months FU visit assessed by TBUT parameter for a Tixel sub-group population only.
Time Frame: Baseline and 6 months post-last treatment (7 months post-baseline)
Population: Tixel sub-group population
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Tixel Group
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
seconds
  Baseline | 4.0 (1.5)
  6 months FU visit | 9.2 (4.0)
  change from baseline - 6 months FU visit | 5.2 (3.8)

12. Other Pre Specified Outcome: Extension Study Endpoint 3
Description: Durability of the clinical benefit effect at 6-months FU visit assessed by MGSS parameter for a Tixel sub-group population only.
Time Frame: Baseline and 6 months post-last treatment (7 months post-baseline)
Population: Tixel sub-group population
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group
Number analyzed (Participants) | 21
Number analyzed (Eyes) | 42
score on a scale
  Baseline | 6.6 (2.3)
  6 months FU visit | 24.8 (10.9)
  change from baseline at 6 months FU visit | 18.2 (10.9)

ADVERSE EVENTS:
Time Frame: 12 months and 10 days
Arm/Group | Tixel Group | LipiFlow
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 4/53 | 1/53
Other Adverse Events (participants affected / at risk) | 6/53 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel Group (N=53) | LipiFlow (N=53)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) — Retinal detachment
Operculated Retinal Hole (Eye disorders) | 1 (1) | 0 (0) — Retinal tear
facial melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — malignant melanoma in situ
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Sepsis
Infectious L5/S1 spondylodiscitis (Infections and infestations) | 1 (1) | 0 (0) — Intervertebral discitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel Group (N=53) | LipiFlow (N=53)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal mass
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) — Bronchitis
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) — COVID-19
Hyprtension (Vascular disorders) | 0 (0) | 1 (1) — Hypetension
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) — Mastoiditis
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Vertigo
Conjunctival cyst (Eye disorders) | 0 (0) | 1 (1) — Conjunctival cyst
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) — Conjunctivitis allergic
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) — Conjunctivitis viral
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Corneal abrasion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT05162261/Prot_SAP_000.pdf